CLINICAL TRIAL: NCT04467879
Title: A Pivotal Study To Evaluate The Effectiveness of Isometric Handgrip Therapy In Prehypertensive And Hypertensive Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New Protocol and Outcome Measures in Review
Sponsor: Zona Health, Inc (Industry)
Collaborators: Research & Development Concierge Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Hypertension, Systolic
Keywords: Diastolic Hypertension; HandGrip Therapy; Pre-Hypertension; Isometric Exercise; Vascular Hypertension
MeSH Terms: conditions — Isolated Systolic Hypertension; Prehypertension; Hypertension

STUDY DESIGN:
Intervention Model Description: Prospective, double-blinded, randomized, sham-controlled study
Who Masked: Participant, Investigator
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Zona Plus - Active - "Normal Grip" (Experimental): Using the Zona Plus Device, the patient will perform a twelve-minute isometric handgrip therapy session at approximately the same time each day . After an initial handgrip strength assessment (the session calibration), a two-minute isometric routine is performed four times, two sessions per hand, with a one-minute non-grip, or rest session between each isometric routine.
  Interventions: Device: Zona Plus Device
- Control Device - Sham - "Weaker Grip" (Sham Comparator): Using the Zona Sham Control Device the patient will perform a twelve-minute isometric handgrip therapy session at approximately the same time each day. After an initial handgrip strength assessment (the calibration), a two-minute isometric routine is performed four times, two sessions per hand, with a one-minute non-grip, or rest session between each isometric routine.
  Interventions: Device: Control Device

INTERVENTIONS:
Device: Zona Plus Device — Zona Plus 3.0 Individualized Isometric Handgrip Therapy Device
  Other Names: Zona Plus 3.0
  Arms: Zona Plus - Active - "Normal Grip"
Device: Control Device — Zona Plus control sham device, with a nominal weaker grip
  Arms: Control Device - Sham - "Weaker Grip"

SUMMARY:
This is a double-blind, sham-controlled clinical trial assessing the effectiveness of personalized isometric handgrip device therapy. Approximately 230 patients who present with a Systolic Blood Pressure reading of ≤ 149mmHg and who have not taken any antihypertensive medication for more than 30 days will be enrolled.

DETAILED DESCRIPTION:
This study is designed to examine the effectiveness of individualized isometric handgrip device therapy in prehypertension or hypertension patient subjects who are not at target BP and who are naive to anti-hypertensive medication for at least 30 days before screening. The investigational plan examines changes in blood pressure (BP) in up to 230 patient subjects who are randomized to either the "active" (i.e., the Zona Plus device proposed for marketing), or to a "sham" device (which is intentionally calibrated for a "weaker grip").

ELIGIBILITY:
Inclusion Criteria

* Male or female of any ethnicity between 18 and 80 years of age
* Diagnosed with prehypertension or hypertension and verified during the Baseline visit
* Non-use of antihypertensive medication for ≥30 prior to screening
* Currently not taking any antihypertensive medications or decline to take any antihypertensive medications(e.g., diuretic, angiotensin-converting enzyme inhibitor (ACEI), angiotensin II receptor blocker (ARB), ] beta-blocker (BB), renin inhibitor (RI), calcium channel blocker (CCB) or alpha-adrenergic agonist (clonidine))
* Sufficient vision with the patient able to see the screen prompts on the device, sufficient hearing with the patient able to hear the device audio prompts, sufficient hand strength (demonstrated by a maximum voluntary contraction equaling 35 units of force in both hands measured by the device)
* Baseline Blood Pressure measurements collected and study device training completed during the Baseline visit
* Non-use of medications and over the counter (OTC)supplement regimen related to hypertension throughout the study duration
* Only one patient per household can participate in the study, eliminating the potential of unblinding
* Able to comply with study procedures and agrees to complete all required study visits and associated activities
* Ability to give written informed consent in either English, Spanish or French •≤149 mmHg, Systolic Blood Pressure wherein patients who present with Systolic Blood Pressure readings ≥140 mmHg will receive heightened monitoring throughout the first month of the study

Exclusion Criteria

* Pregnant or not using adequate contraception
* Blood Pressure ≥150 mmHg (systolic) and/or >90 mmHg (diastolic)
* History of heart failure
* Hospitalization due to a hypertensive emergency, with impending or progressive target organ dysfunction (i.e., renal dysfunction, left ventricular hypertrophy or CNS involvement) within the past six (6) months

  •>10 mmHg difference in Systolic Blood Pressure between the right and left arms collected during screening
* Unstable Blood Pressure, defined as >5 mmHg variance between any two (2) consecutive weekly readings (with a maximum of four (4) attempts) to determine a baseline BP measurement
* Arm circumference greater than 45cm
* Acute illness, infection, or inflammation
* Unstable cardiovascular disorder, such as MI, unstable angina, significant arrhythmia, stroke, or TIA within the last six (6)months, or other serious comorbidity impacting life expectancy to < than a 1 year
* Rest or exertional angina pectoris in the previous six (6) months
* History of solid organ transplant
* Secondary form of hypertension (HTN) etiology, including but not limited to primary aldosteronism, chronic steroid therapy and Cushing syndrome, pheochromocytoma, aorta coarctation or untreated thyroid or parathyroid disease
* Concurrent participation in an investigational clinical study that has not completed the follow-up period or planned participation in another study within the next six(6) months
* Any condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete, good quality data or the completion of the research study
* Currently own or have owned another Zona Plus device and are,or have been,voluntarily performing the isometric handgrip activities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Systolic Blood Pressure to Day 70 ± 2 Days | Change from Baseline to Day 70 ±2 Days
  Comparative assessment in the change from Baseline in seated cuff Systolic Blood Pressure after ten(10) weeks of treatment between patients treated with the Zona Plus nominal device ("stronger grip") and patients treated with the Placebo control device ("weaker grip"). A reduction in Systolic Blood ≥ 5 Preassure after 10 weeks of treatment is considered to be a better outcome.

SECONDARY OUTCOMES:
Change from Baseline in Diastolic Blood Pressure to Day 70 ± 2 Days | Change from Baseline to Day 70 ±2 Days
  Comparative assessment of the change from Baseline in seated cuff Diastolic Blood Pressure after 10 weeks of treatment between patients treated with the Zona Plus nominal device ("stronger grip") and patients treated with the Placebo control device ("weaker grip").
Percentage change from Baseline in Systolic Blood Pressure reduction at Day 70 ± 2 Days | Change from Baseline to Day 70 ± 2 Days
  Comparative assessment in the percentage of patients who achieve a clinically significant Systolic Blood Pressure reduction (defined as ≥ 5 mmHg) at Day 70 ± 2 Days.
Percentage change from Baseline in Diastolic Blood Pressure reduction at Day 70 ± 2 Days | Change from Baseline to Day 70 ± 2 Days
  Comparative assessment in the percentage of patients who achieve a clinically significant Diastolic Blood Pressure reduction (defined as ≥3 mmHg) at Day 70 ± 2 Days.
Percentage change from Baseline in Systolic Blood Pressure reduction at Day 160 ± 4 Days | Change from Baseline to Day 160 ± 4 Days
  Comparative assessment in change from Baseline in the seated cuff Systolic Blood Pressure after 6 months Day 160 ± 4 of treatment between patients treated with the Zona Plus nominal device and patients treated with the Placebo control device.
Percentage change in Diastolic Blood Pressure reduction at Day 160 ± 4 Days | Change from Baseline to Day 160 ± 4 Days
  Comparative assessment in change from Baseline in the seated cuff Diastolic Blood Pressure after 6 months Day 160 ± 4 Days of treatment between patients treated with the Zona Plus nominal device and patients treated with the Placebo control device.
Percentage change from Baseline in Systolic Blood Pressure reduction at Day 160 ± 4 Days | Change from Baseline to Day 160 ± 4 Days
  Comparative assessment in the percentage of patients who achieve a clinically significant Systolic Blood Pressure reduction (defined as ≥ 5 mmHg) at Day 160 ± 4 Days
Percentage change in Diastolic Blood Pressure reduction at Day 160 ± 4 Days | Change from Baseline to Day 160 ± 4 Days
  Comparative assessment in the percentage of patients who achieve a clinically significant Diastolic Blood Pressure reduction defined as ≥3 mmHg at Day 160 ± 4 Days
Comparison of Heart Rate between Zona Plus nominal device and Placebo controlled device | Change from Baseline to Day 160 ± 4 Days
  The Heart Rate (HR) will be recorded and compared between the Zona Plus nominal device and the Placebo control device treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Young, Study Chair — Zona Health, Inc
Locations (5):
- United States (5):
  - Saint Louis Heart & Vascular, P.C., St Louis, Missouri
  - Carolinas Research Center LLC, Charlotte, North Carolina
  - Goldsboro Medical Center, Goldsboro, North Carolina
  - Sante Clinical Research, Kerrville, Texas
  - Sun Research Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
If in the future Investigators want to access the data for secondary analysis they can submit a request from the Sponsor or R&D Data Management Contact. Individual patient data will not be shared by the sponsor directly and will be aggregated, monitored, and de-identified (APD) via 1) final approved clinical study report 2) any manuscripts or summary results report via an email request to the central contact once database lock has occurred and reports are generated.

REFERENCES:
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Al-Khatib SM, Califf RM, Hasselblad V, Alexander JH, McCrory DC, Sugarman J. Medicine. Placebo-controls in short-term clinical trials of hypertension. Science. 2001 Jun 15;292(5524):2013-5. doi: 10.1126/science.1057783. No abstract available. PMID 11408643
- [Background] ALLHAT Officers and Coordinators for the ALLHAT Collaborative Research Group. The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. Major outcomes in high-risk hypertensive patients randomized to angiotensin-converting enzyme inhibitor or calcium channel blocker vs diuretic: The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). JAMA. 2002 Dec 18;288(23):2981-97. doi: 10.1001/jama.288.23.2981. PMID 12479763
- [Background] Bakke EF, Hisdal J, Kroese AJ, Jorgensen JJ, Stranden E. Blood pressure response to isometric exercise in patients with peripheral atherosclerotic disease. Clin Physiol Funct Imaging. 2007 Mar;27(2):109-15. doi: 10.1111/j.1475-097X.2007.00720.x. PMID 17309531
- [Background] Balasubramanian V, Mann S, Millar-Craig MW, Raftery EB. Effect of labetalol in hypertension during exercise and postural changes. Br J Clin Pharmacol. 1979 Apr;8 Suppl 2:95S-100S. doi: 10.1111/j.1365-2125.1979.tb04761.x. PMID 26635176
- [Background] Black HR, Elliott WJ, Neaton JD, Grandits G, Grambsch P, Grimm RH Jr, Hansson L, Lacouciere Y, Muller J, Sleight P, Weber MA, White WB, Williams G, Wittes J, Zanchetti A, Fakouhi TD, Anders RJ. Baseline Characteristics and Early Blood Pressure Control in the CONVINCE Trial. Hypertension. 2001 Jan;37(1):12-18. doi: 10.1161/01.hyp.37.1.12. PMID 11208750
- [Background] Boutcher SH, Stocker D. Cardiovascular responses to light isometric and aerobic exercise in 21- and 59-year-old males. Eur J Appl Physiol Occup Physiol. 1999 Aug;80(3):220-6. doi: 10.1007/s004210050585. PMID 10453924
- [Background] Buck C, Donner AP. Isometric occupational exercise and the incidence of hypertension. J Occup Med. 1985 May;27(5):370-2. doi: 10.1097/00043764-198505000-00017. PMID 4009307
- [Background] Chrysant SG. Current evidence on the hemodynamic and blood pressure effects of isometric exercise in normotensive and hypertensive persons. J Clin Hypertens (Greenwich). 2010 Sep;12(9):721-6. doi: 10.1111/j.1751-7176.2010.00328.x. PMID 20883233
- [Background] Cushman WC, Ford CE, Cutler JA, Margolis KL, Davis BR, Grimm RH, Black HR, Hamilton BP, Holland J, Nwachuku C, Papademetriou V, Probstfield J, Wright JT Jr, Alderman MH, Weiss RJ, Piller L, Bettencourt J, Walsh SM; ALLHAT Collaborative Research Group. Success and predictors of blood pressure control in diverse North American settings: the antihypertensive and lipid-lowering treatment to prevent heart attack trial (ALLHAT). J Clin Hypertens (Greenwich). 2002 Nov-Dec;4(6):393-404. doi: 10.1111/j.1524-6175.2002.02045.x. PMID 12461301
- [Background] Eguchi K, Yacoub M, Jhalani J, Gerin W, Schwartz JE, Pickering TG. Consistency of blood pressure differences between the left and right arms. Arch Intern Med. 2007 Feb 26;167(4):388-93. doi: 10.1001/archinte.167.4.388. PMID 17325301
- [Background] Fotherby MD, Panayiotou B, Potter JF. Age-related differences in simultaneous interarm blood pressure measurements. Postgrad Med J. 1993 Mar;69(809):194-6. doi: 10.1136/pgmj.69.809.194. PMID 8497433
- [Background] Gasowski J, Staessen JA, Celis H, Fagard RH, Thijs L, Birkenhager WH, Bulpitt CJ, Fletcher AE, Arabidze GG, de Leeuw P, Dollery CT, Duggan J, Kawecka-Jaszcz K, Leonetti G, Nachev C, Safar M, Rodico JL, Rosenfeld J, Seux ML, Tuomilehto J, Webster J, Yodfat Y. Systolic Hypertension in Europe (Syst-Eur) trial phase 2: objectives, protocol, and initial progress. Systolic Hypertension in Europe Investigators. J Hum Hypertens. 1999 Feb;13(2):135-45. doi: 10.1038/sj.jhh.1000769. PMID 10100063
- [Background] Grucza R, Kahn JF, Cybulski G, Niewiadomski W, Stupnicka E, Nazar K. Cardiovascular and sympatho-adrenal responses to static handgrip performed with one and two hands. Eur J Appl Physiol Occup Physiol. 1989;59(3):184-8. doi: 10.1007/BF02386185. PMID 2583160
- [Background] Hansson L, Zanchetti A, Carruthers SG, Dahlof B, Elmfeldt D, Julius S, Menard J, Rahn KH, Wedel H, Westerling S. Effects of intensive blood-pressure lowering and low-dose aspirin in patients with hypertension: principal results of the Hypertension Optimal Treatment (HOT) randomised trial. HOT Study Group. Lancet. 1998 Jun 13;351(9118):1755-62. doi: 10.1016/s0140-6736(98)04311-6. PMID 9635947
- [Background] Howden R, Lightfoot JT, Brown SJ, Swaine IL. The effects of isometric exercise training on resting blood pressure and orthostatic tolerance in humans. Exp Physiol. 2002 Jul;87(4):507-15. doi: 10.1111/j.1469-445x.2002.tb00064.x. PMID 12392115
- [Background] Hurst JW, Morris DC, Alexander RW. The use of the New York Heart Association's classification of cardiovascular disease as part of the patient's complete Problem List. Clin Cardiol. 1999 Jun;22(6):385-90. doi: 10.1002/clc.4960220604. PMID 10376176
- [Background] Julius S, Kjeldsen SE, Weber M, Brunner HR, Ekman S, Hansson L, Hua T, Laragh J, McInnes GT, Mitchell L, Plat F, Schork A, Smith B, Zanchetti A; VALUE trial group. Outcomes in hypertensive patients at high cardiovascular risk treated with regimens based on valsartan or amlodipine: the VALUE randomised trial. Lancet. 2004 Jun 19;363(9426):2022-31. doi: 10.1016/S0140-6736(04)16451-9. PMID 15207952
- [Background] Kelley GA, Kelley KS. Isometric handgrip exercise and resting blood pressure: a meta-analysis of randomized controlled trials. J Hypertens. 2010 Mar;28(3):411-8. doi: 10.1097/HJH.0b013e3283357d16. PMID 20009767
- [Background] Kerber RE, Miller RA, Najjar SM. Myocardial ischemic effects of isometric, dynamic and combined exercise in coronary artery disease. Chest. 1975 Apr;67(4):388-94. doi: 10.1378/chest.67.4.388. PMID 1122766
- [Background] Lewis SF, Taylor WF, Bastian BC, Graham RM, Pettinger WA, Blomqvist CG. Haemodynamic responses to static and dynamic handgrip before and after autonomic blockade. Clin Sci (Lond). 1983 Jun;64(6):593-9. doi: 10.1042/cs0640593. PMID 6839666
- [Background] McGowan CL, Levy AS, Millar PJ, Guzman JC, Morillo CA, McCartney N, Macdonald MJ. Acute vascular responses to isometric handgrip exercise and effects of training in persons medicated for hypertension. Am J Physiol Heart Circ Physiol. 2006 Oct;291(4):H1797-802. doi: 10.1152/ajpheart.01113.2005. Epub 2006 Apr 28. PMID 16648182
- [Background] McGowan CL, Visocchi A, Faulkner M, Verduyn R, Rakobowchuk M, Levy AS, McCartney N, MacDonald MJ. Isometric handgrip training improves local flow-mediated dilation in medicated hypertensives. Eur J Appl Physiol. 2007 Feb;99(3):227-34. doi: 10.1007/s00421-006-0337-z. Epub 2006 Nov 15. PMID 17106718
- [Background] Millar PJ, Bray SR, McGowan CL, MacDonald MJ, McCartney N. Effects of isometric handgrip training among people medicated for hypertension: a multilevel analysis. Blood Press Monit. 2007 Oct;12(5):307-14. doi: 10.1097/MBP.0b013e3282cb05db. PMID 17890969
- [Background] Millar PJ, Bray SR, MacDonald MJ, McCartney N. The hypotensive effects of isometric handgrip training using an inexpensive spring handgrip training device. J Cardiopulm Rehabil Prev. 2008 May-Jun;28(3):203-7. doi: 10.1097/01.HCR.0000320073.66223.a7. PMID 18496321
- [Background] Millar PJ, MacDonald MJ, Bray SR, McCartney N. Isometric handgrip exercise improves acute neurocardiac regulation. Eur J Appl Physiol. 2009 Nov;107(5):509-15. doi: 10.1007/s00421-009-1142-2. Epub 2009 Aug 13. PMID 19680681
- [Background] Millar PJ, MacDonald MJ, McCartney N. Effects of isometric handgrip protocol on blood pressure and neurocardiac modulation. Int J Sports Med. 2011 Mar;32(3):174-80. doi: 10.1055/s-0030-1268473. Epub 2010 Dec 16. PMID 21165806
- [Background] Murakami E, Matsuzaki K, Sumimoto T, Mukai M, Kazatani Y, Kodama K. Clinical significance of pressor responses to laboratory stressor testing in hypertension. Hypertens Res. 1996 Jun;19(2):133-7. doi: 10.1291/hypres.19.133. PMID 10968206
- [Background] Owen A, Wiles J, Swaine I. Effect of isometric exercise on resting blood pressure: a meta analysis. J Hum Hypertens. 2010 Dec;24(12):796-800. doi: 10.1038/jhh.2010.13. Epub 2010 Feb 25. PMID 20182455
- [Background] Peters PG, Alessio HM, Hagerman AE, Ashton T, Nagy S, Wiley RL. Short-term isometric exercise reduces systolic blood pressure in hypertensive adults: possible role of reactive oxygen species. Int J Cardiol. 2006 Jun 16;110(2):199-205. doi: 10.1016/j.ijcard.2005.07.035. Epub 2005 Oct 18. PMID 16239039
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ. Recommendations for blood pressure measurement in humans and experimental animals: part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Circulation. 2005 Feb 8;111(5):697-716. doi: 10.1161/01.CIR.0000154900.76284.F6. PMID 15699287
- [Background] Ray CA, Carrasco DI. Isometric handgrip training reduces arterial pressure at rest without changes in sympathetic nerve activity. Am J Physiol Heart Circ Physiol. 2000 Jul;279(1):H245-9. doi: 10.1152/ajpheart.2000.279.1.H245. PMID 10899063
- [Background] Rosenthal T, Oparil S. Hypertension in women. J Hum Hypertens. 2000 Oct-Nov;14(10-11):691-704. doi: 10.1038/sj.jhh.1001095. PMID 11095160
- [Background] Sacks FM, Svetkey LP, Vollmer WM, Appel LJ, Bray GA, Harsha D, Obarzanek E, Conlin PR, Miller ER 3rd, Simons-Morton DG, Karanja N, Lin PH; DASH-Sodium Collaborative Research Group. Effects on blood pressure of reduced dietary sodium and the Dietary Approaches to Stop Hypertension (DASH) diet. DASH-Sodium Collaborative Research Group. N Engl J Med. 2001 Jan 4;344(1):3-10. doi: 10.1056/NEJM200101043440101. PMID 11136953
- [Background] Prevention of stroke by antihypertensive drug treatment in older persons with isolated systolic hypertension. Final results of the Systolic Hypertension in the Elderly Program (SHEP). SHEP Cooperative Research Group. JAMA. 1991 Jun 26;265(24):3255-64. PMID 2046107
- [Background] Taylor AC, McCartney N, Kamath MV, Wiley RL. Isometric training lowers resting blood pressure and modulates autonomic control. Med Sci Sports Exerc. 2003 Feb;35(2):251-6. doi: 10.1249/01.MSS.0000048725.15026.B5. PMID 12569213
- [Background] Whelton PK, He J, Appel LJ, Cutler JA, Havas S, Kotchen TA, Roccella EJ, Stout R, Vallbona C, Winston MC, Karimbakas J; National High Blood Pressure Education Program Coordinating Committee. Primary prevention of hypertension: clinical and public health advisory from The National High Blood Pressure Education Program. JAMA. 2002 Oct 16;288(15):1882-8. doi: 10.1001/jama.288.15.1882. PMID 12377087
- [Background] Badrov MB, Freeman SR, Zokvic MA, Millar PJ, McGowan CL. Isometric exercise training lowers resting blood pressure and improves local brachial artery flow-mediated dilation equally in men and women. Eur J Appl Physiol. 2016 Jul;116(7):1289-96. doi: 10.1007/s00421-016-3366-2. Epub 2016 May 2. PMID 27137950
- [Background] Wiley RL, Dunn CL, Cox RH, Hueppchen NA, Scott MS. Isometric exercise training lowers resting blood pressure. Med Sci Sports Exerc. 1992 Jul;24(7):749-54. PMID 1501558
- [Background] Division of Cardiovascular and Renal Drug Products, Center for Drug Evaluation andResearch (CDER), Food,and Drug Administration. Guidance forIndustry.Hypertension Indication: Drug Labeling for Cardiovascular Outcome Claims. 2008.http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatorylnformation/Guidances/ucm075072.pdf
- [Background] Gibbons RJ, Balady GJ, Bricker JT, Chaitman BR, Fletcher GF, Froelicher VF, Mark DB, McCallister BD, Mooss AN, O'Reilly MG, Winters WL Jr, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Russell RO, Smith SC Jr; American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1997 Exercise Testing Guidelines). ACC/AHA 2002 guideline update for exercise testing: summary article: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1997 Exercise Testing Guidelines). Circulation. 2002 Oct 1;106(14):1883-92. doi: 10.1161/01.cir.0000034670.06526.15. No abstract available. PMID 12356646
- [Background] Hicks KA, Hung HMJ, Mahaffey KW, et al.
- [Background] ICH Steering Committee. Draft ICH Consensus Principle:Principles for ClinicalEvaluation ofNew Antihypertensive Drugs. International Conference onHarmonisation ofTechnical Requirements for Registration of Pharmaceuticals forHuman Use. 2000.http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/ucm073147.pdf
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Kiveloff B, Huber O. Brief maximal isometric exercise in hypertension. J Am Geriatr Soc. 1971 Dec;19(12):1006-12. doi: 10.1111/j.1532-5415.1971.tb02221.x. No abstract available. PMID 5153689
- [Background] Millar, PJ. Isometric handgrip training: a natural hypertensive therapy. TownsendLetter: The Examiner of Alternative Medicine 2008.
- [Background] Millar PJ, Paashuis A, McCartney. Isometric Handgrip Effects on Hypertension. CurrHypertens Rev 2009;5:54-60
- See also: Drug Labeling for Cardiovascular Outcome Claims — http://www.fda.gov/regulatory-information/search-fda-guidance-documents/hypertension-indication-drug-labeling-cardiovascular-outcome-claims
- See also: Principles for ClinicalEvaluation ofNew Antihypertensive Drugs. — http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/ucm073147.pdf
- See also: The Seventh Report of the Joint National Committee on Prevention, Detection,Evaluation, and Treatment of High Blood Pressure — http://www.nhlbi.nih.gov/files/docs/guidelines/jnc7full.pdf